CLINICAL TRIAL: NCT06737393
Title: Postoperative Bladder Filling After Outpatient Laparoscopic Hysterectomy and Time to Discharge: a Randomized Controlled Trial
Brief Title: Postoperative Bladder Filling After Outpatient Laparoscopic Hysterectomy and Time to Discharge
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-09979-FB
Record Dates: First submitted 2024-07-15; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-07

CONDITIONS: Patient Discharge; Urinary Complication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Backfill (Experimental): Participants will receive 200 mL of room temperature, sterile normal saline instilled retrograde into the bladder at the completion of the surgery prior to Foley catheter removal and the Foley subsequently removed intraoperatively.
  Interventions: Procedure: Backfill
- No bladder filling (No Intervention): Participants will have the Foley catheter removed intraoperatively at completion of the procedure.

INTERVENTIONS:
Procedure: Backfill — Participants undergoing laparoscopic hysterectomy have the bladder filled with 200 mL saline prior to Foley removal at the end of surgery.
  Arms: Backfill

SUMMARY:
The investigators hypothesize that backfilling the bladder postoperatively will reduce time to spontaneous void and subsequent discharge from the post-anesthesia care unit.

DETAILED DESCRIPTION:
This is a prospective, single-blinded, randomized clinical trials in which patients undergoing laparoscopic hysterectomy will be randomized in a 1:1 ratio to have the bladder backfilled at the completion of the surgery prior to Foley catheter removal. If the patient is assigned to group A, 200 mL of room temperature, sterile normal saline will be instilled retrograde into the bladder at the completion of the surgery prior to Foley catheter removal and the Foley subsequently removed intraoperatively. If the patient is assigned to group B, the Foley catheter will be removed intraoperatively at completion of the procedure. The standard protocol is to use a 16F Foley catheter for gynecologic laparoscopy cases, and patients in both groups will receive the same size catheter. After surgery, time to discharge and time to void will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 80
* Undergoing planned laparoscopic hysterectomy as a day surgery procedure

Exclusion Criteria:

* Women younger than 18 or older than 80 years of age
* Undergoing a non-laparoscopic unplanned surgical procedure

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who are biologically female
Enrollment: 112 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Time to discharge | Within 3 days following surgery
  The time to discharge for each participant, which will be defined as the length of time from surgery completion to discharge from the post-anesthesia care unit, will be recorded.

SECONDARY OUTCOMES:
Time to void | Within 3 days following surgery
  The time to void for each participant, which will be defined as the length of time from surgery completion to the time of participant's first voiding event, will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chao L, Mansuria S. Postoperative Bladder Filling After Outpatient Laparoscopic Hysterectomy and Time to Discharge: A Randomized Controlled Trial. Obstet Gynecol. 2019 May;133(5):879-887. doi: 10.1097/AOG.0000000000003191. PMID 30969209
- [Background] Ghezzi F, Cromi A, Uccella S, Colombo G, Salvatore S, Tomera S, Bolis P. Immediate Foley removal after laparoscopic and vaginal hysterectomy: determinants of postoperative urinary retention. J Minim Invasive Gynecol. 2007 Nov-Dec;14(6):706-11. doi: 10.1016/j.jmig.2007.06.013. PMID 17980330
- [Background] Du J, Marshall D, Leyland J, Shaw L, Broome KE, Mason DF. Prospective, multicentre, randomized controlled trial of bladder filling prior to trial of void on the timing of discharge. ANZ J Surg. 2013 Apr;83(4):239-42. doi: 10.1111/j.1445-2197.2012.06253.x. Epub 2012 Sep 18. PMID 22984818
- [Background] Hariati H, Suza DE, Tarigan R. Risk Factors Analysis for Catheter-Associated Urinary Tract Infection in Medan, Indonesia. Open Access Maced J Med Sci. 2019 Sep 12;7(19):3189-3194. doi: 10.3889/oamjms.2019.798. eCollection 2019 Oct 15. PMID 31949514

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT06737393/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT06737393/ICF_001.pdf